CLINICAL TRIAL: NCT04141150
Title: A Phase 2, Multicenter Study of [18F]APN-1607 Positron Emission Tomography in Subjects With Alzheimer's Disease Compared to Healthy Subjects
Brief Title: Evaluation of [18F]APN-1607 PET Uptake in Alzheimer's Disease Patients Compared With Healthy Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: APRINOIA Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Organization: APRINOIA Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APN-1607-201
Record Dates: First submitted 2019-10-17; First posted 2019-10-28 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment Due to Alzheimer's Disease; Healthy Volunteers
Keywords: AD; MDAD; HV
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]APN-1607 (Experimental): Subjects will undergo PET imaging using [18F]APN-1607.
  Interventions: Drug: [18F]APN-1607

INTERVENTIONS:
Drug: [18F]APN-1607 — In this study, all patients will receive one injection of [18F]APN-1607, a PET radiopharmaceutical selective for fibrillar tau. For the injection, subjects will receive a target dose of 7 mCi IV as a bolus injection. [18F]APN-1607 injection will be followed by a 10 ml saline flush.

SUMMARY:
The overall objective of this study is to compare the overall pattern of [18F]APN-1607 uptake in subjects with MDAD, subjects with AD dementia, and healthy subjects.

DETAILED DESCRIPTION:
The overall objective of this study is to compare the overall pattern of [18F]APN-1607 uptake in subjects with MDAD, subjects with AD dementia, and healthy subjects.

The specific objectives are:

* To expand the safety and tolerability profile for the administration of [18F]APN-1607 and PET scanning.
* To assess regional patterns of [18F]APN-1607 uptake.
* To determine the Braak stage equivalent reflected by [18F]APN-1607 uptake patterns.
* To evaluate the relationship between regional measures of [18F]APN-1607 uptake and demographic characteristics, eg, age and gender; biological characteristics, eg, apolipoprotein E epsilon 4 (APOE4) carrier status and measures of Aβ burden; and clinical characteristics, eg, measurements of AD disease severity, such as National Institute on Aging and Alzheimer's Association (NIA-AA) diagnosis, Mini-mental Status Exam (MMSE) score, and Alzheimer's Disease Assessment Scale-cognitive subscale (ADAScog).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for All Subjects:

1. Males or females aged 50 to 85 years, inclusive.
2. Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year (ie, 12 consecutive months with no menses without an alternative medical cause) or, if they are of childbearing potential, must commit to using a barrier contraception method or to abstinence for the duration of the study and must have a negative pregnancy test.
3. Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method (ie, condom), or to abstinence for the study duration.
4. Male subjects must not donate sperm for the study duration.
5. Willing and able to participate in all study procedures.

Additional Inclusion Criteria for Healthy Subjects:

1. Written informed consent must be obtained before any assessment is performed.
2. Medically healthy with no clinically relevant finding on physical examination, laboratory profiles, VS, or ECG at screening and upon reporting for the [18F]APN-1607 Imaging Visit.
3. No cognitive impairment based on neuropsychological battery and as judged by the Investigator.
4. No first-degree family history of early-onset AD or other neurodegenerative disease associated with dementia (prior to age 65).
5. Has a clinical dementia rating (CDR) score of 0.
6. Has an MMSE score ≥ 27.
7. The subject has an appropriate informant to accompany the subject to screening to provide information for the CDR testing. In the event that the informant cannot accompany the subject to screening, the interview may be performed via phone, at the discretion of the site Investigator.

Additional Inclusion Criteria for Subjects with MDAD:

1. Written informed consent must be obtained before any assessment is performed.
2. Must meet all of the clinical criteria for MCI according to NIA-AA criteria, including lack of functional impairment sufficient to warrant a diagnosis of dementia.
3. Has a CDR score = 0.5.
4. Has an MMSE score between 24 and 30, inclusive.
5. Has a positive amyloid PET scan obtained during screening or in the past 1 year.
6. Medications taken for symptomatic treatment of AD must have been stable for at least 30 days prior to screening and throughout the completion of the neuropsychological battery.
7. The subject has an appropriate informant to provide information for the CDR and accompany the subject for any visits, if required for subject or staff comfort or safety.

Additional Inclusion Criteria for Subjects with AD Dementia:

1. Written informed consent must be obtained before any assessment is performed. If in the Investigator's opinion the subject lacks capacity to consent, participation is only possible if the subject has a legally authorized representative (LAR) or responsible next-of-kin and that individual provides written informed consent in accordance with local regulations and guidelines and the rules of the applicable independent ethics committee (IEC)/institutional review board (IRB). When written informed consent is provided by a LAR or responsible next of kin, the subject's assent must also be obtained and documented. For subjects judged lacking capacity to consent, next-of-kin consent in lieu of LAR consent is only allowed where permitted by local laws and regulations.
2. Has a diagnosis of AD dementia according to NIA-AA criteria, including significant impairment of activities of daily living.
3. Has a CDR score ≥ 0.5 at screening.
4. Has an MMSE score between 10 and 26, inclusive.
5. Has a positive amyloid PET scan obtained during screening or in the past 1 year.
6. Medications taken for symptomatic treatment of AD must have been stable for 30 days prior to screening and throughout the completion of the neuropsychological battery.
7. The subject has an appropriate informant to accompany the subject on all visits and provide information for the CDR.

Exclusion Criteria for All Subjects:

1. Current or prior history (within the last 10 years) of alcohol or drug abuse.
2. Known hypersensitivity to [18F]APN-1607 or its excipients
3. Clinically significant active or unstable medical illness or planned surgical procedures during the study period. History of cancer (other than non-melanoma skin cancers or stable, local prostate cancer), unless without evidence of active disease within the last 3 years and without ongoing medical or surgical therapy.
4. Laboratory tests with clinically significant abnormalities or a history or evidence of clinically significant unstable medical illness.
5. Has received any investigational drug or device for any purpose within 30 days of screening (or 5 halflives of the drug, whichever is longer), has received a non-biologic investigational treatment (ie, small molecule) for AD or other cause of dementia within the last 3 months (or 5 half-lives of the drug, whichever is longer), or received a non-vaccine treatment (ie, monoclonal antibody) for the treatment of AD or other cause of dementia within the last 6 months, or has ever received a vaccine for the treatment of AD or other cause of dementia.
6. Prior participation in other research protocols or clinical care in the last year in which the additional radiation exposure expected from participation in this clinical study will together exceed local guidelines, eg, above an effective dose of 50 mSv in the US.
7. Pregnant, lactating or breastfeeding.
8. Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
9. Unsuitable veins for repeated venipuncture.
10. MRI exclusion criteria include: Findings that may be responsible for the neurologic status of the patient such as significant evidence of cerebrovascular disease (more than two lacunar infarcts, any territorial infarct >1cm3, or deep white matter abnormality corresponding to an overall Fazekas scale of 3 with at least one confluent hyperintense lesion on the fluid-attenuated inversion recovery (FLAIR) sequence that is ≥20 mm in any dimension), infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with central nervous system (CNS) disease. For subjects with MDAD or AD dementia, there may be evidence of atrophy compatible with AD.
11. Implants, such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI unless an acceptable MRI obtained in the 1 year prior to participation in the study is used.
12. Signs or symptoms suggestive of active Coronavirus disease 2019 (COVID-19) and/or confirmed diagnosis of COVID-19, or positive COVID-19 polymerase chain reaction (PCR) test in the previous 2 weeks. These subjects should not be enrolled until 4 weeks after full recovery and further assessment by the Investigator per institutional guidelines. A subject with a known history of being exposed to someone who was diagnosed of COVID-19, during the prior 4 weeks, should not be enrolled unless the infection is excluded by local practice or institution.

Exclusion Criteria for Healthy Subjects:

1. Meets criteria for a diagnosis of MDAD or dementia or has ever had such a diagnosis.
2. Has ever received treatment with a drug for cognitive impairment or dementia.

Exclusion Criteria for Subjects with MDAD:

1. Meets criteria for a diagnosis of dementia due to AD.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of [18F]APN-1607 Uptake Patterns by Regional SUVR Values | Day 7
  Regional [18F]APN-1607 uptake patterns will be assessed in regions of interest (ROIs) and an iROI that are relevant to AD pathology. [18F]APN-1607 uptake patterns identified by regional analysis will be compared among healthy subjects, subjects with MDAD, and subjects with AD dementia. Standard uptake value (SUV) will be calculated for each ROI, and SUVRs will be calculated by normalizing SUV of ROIs to the SUV of relevant reference region. Mean and standard deviation of [18F]APN-1607 uptake (ie, SUVR) will be calculated across healthy, MDAD and AD dementia cohorts. Differences between groups will be tested at a P-value of 0.05 using statistical analyses methods (eg, unpaired t-test, ANOVA).

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | Day 7
  Measured by participants reporting AEs through non-directive questioning of the subject at each visit during the study or when volunteered by participants during or between visits.
Number of Serious Adverse Events (SAEs) | Day 7
  Measured by participants reporting adverse events classified as serious
Number of participants with vital sign abnormalities | Day 7
  Vital Sign measurements will include blood pressure, pulse rate, respiratory rate and body temperature.
Number of participants with ECG abnormalities | Day 7
  Measured by 12-lead electrocardiogram
Number of participants with clinical laboratory abnormalities | Day 7
  Measured by blood and urine analysis

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, M.D., Ph.D, Principal Investigator — Invicro
Locations (3):
- United States (3):
  - Invicro (Site 100), 60 Temple Street, 8th Floor, New Haven, Connecticut
  - The NeuroCognitive Institute (Site 103), 111 Howard Blvd., Suite 204, Mount Arlington, New Jersey
  - Columbia University Irving Center for Clinical and Translational Research (Site 105), 622 West 168th Street, PH-10th Floor, New York, New York

REFERENCES:
- See also: Description Related Information — https://invicro.com